CLINICAL TRIAL: NCT06704243
Title: Peer Support Group for AYA Allogeneic Stem Cell Transplant Recipients
Brief Title: Peer Support Group for Adolescent and Young Adult (AYA) Allogeneic Stem Cell Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Samantha Mayo, Clinician Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5959
Record Dates: First submitted 2024-10-25; First posted 2024-11-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Leukemia; Stem Cell Transplant
Keywords: peer support; adolescents and young adults
MeSH Terms: conditions — Neoplasms; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Support (Experimental): The intervention will be a monthly online AYA peer support group (1 hour) that will run for six months via Microsoft Teams.
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Peer Support — The intervention will be a monthly online AYA peer support group (1 hour) that will run for six months via Microsoft Teams.
  In an effort to evaluate a patient-driven "real-world" intervention, the support group has been designed with the following features: 1) participants will be asked to commit for a six month period, but are able to miss sessions if necessary; and, 2) each session will be facilitated by a Nurse Practitioner and Social Worker from the Allo-HSCT program, but the topics of discussion will be determined by the AYA participants present at each session. Participants in the group will then be invited to share their thoughts and experiences about these topics, with as much information as they feel comfortable.

SUMMARY:
Allogeneic Haemopoietic Stem Cell Transplant (Allo-HSCT) is a potentially curative option for patients with both malignant and non-malignant hematological disorders. There appears to be unique experiences that adolescents and young adults (AYA) face when undergoing transplant. There is literature to suggest that peer support for young adults is associated with improvements in mental health including greater happiness, self-esteem and effective coping, as well as reductions in depression, loneliness and anxiety.

Our primary objective is to determine the feasibility and acceptability of an AYA peer support program for patients undergoing Allo-HSCT. Our secondary objective is to explore the impact of the AYA peer support program on sense of support/connectivity, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years of age
* >3 months post Allo-HSCT
* any malignant /non-malignant indication for Allo-HSCT

Exclusion Criteria:

- Non-English speaking

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | at 6 months
  The Feasibility of Intervention Measure (FIM) revised to evaluated the AYA peer support program comprises 4-items regarding the respondent's perceptions of the feasibility of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater feasibility of the intervention.
Acceptability of Intervention Measure (AIM) | at 6 months
  The Acceptability of Intervention Measure (AIM) revised to evaluated the AYA peer support program comprises 4-items regarding the respondent's perceptions of the acceptability of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | at 6 months
  The Intervention Appropriate Measure (IAM) revised to evaluated the AYA peer support program comprises 4-items regarding the respondent's perceptions of the appropriateness of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater appropriateness of the intervention.
Post-intervention Qualitative interviews | at 6 months
  Post-intervention qualitative interviews with participants will also explore their perceptions of the feasibility and acceptability of the intervention, including suggestions for improvement of the intervention. These semi-structured interviews will also help explore participant's opinions related to program length, time, usefulness, and delivery.
Intervention usage | at 6 months
  Intervention usage (i.e. proportion of sessions attended by each participant) will be calculated based on attendance lists for each session collected by the session facilitators. Reasons for non-attendance or early drop-out from a session will be collected, but this is optional for participants.

SECONDARY OUTCOMES:
Social Connectedness | Baseline, 3 months, and 6 months
  The Social Connectedness Scale is a measure of one's sense of belonging or connectedness between the self and other people, including friends and society. It comprises 20-items about one's view of themselves, rated from 1 (strongly disagree) to 6 (strongly agree). Scores are calculated by summing responses to the 20 items. Possible scores range from 20-120, with higher scores indicating better social connectedness.
Anxiety | Baseline, 3 months, and 6 months
  GAD-7 (Generalized Anxiety Disorder screener) is a measure of anxiety. It comprises 7-items about one's bother with anxiety symptoms, rated from 0 (not at all) to 3 (nearly every day). Scores are calculated by summing responses to the 7 items. Possible scores range from 0-21, with higher scores indicating worse anxiety.
Depressive Symptoms | Baseline, 3 months, and 6 months
  PHQ-9 (Patient Health Questionnaire -9) is a measure of depressive symptoms. It comprises 9-items about one's bother with depressive symptoms, rated from 0 (not at all) to 3 (nearly every day). Scores are calculated by summing responses to the 9 items. Possible scores range from 0-27, with higher scores indicating worse depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Mayo, RN PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lee, R. M., Robbins, S. B., & Hill, C. E. (1995). Measuring Belongingness: The Social Connectedness and the Social Assurance Scales. Journal of Counseling Psychology, 42(2), 232-241. https://doi.org/10.1037/0022-0167.42.2.232